CLINICAL TRIAL: NCT01148264
Title: Efficacy of Olanzapine in Break-through Emesis After Prophylaxis With Dexamethasone, 5-HT3 Receptor Antagonists and Aprepitant Compared to Metoclopramide
Brief Title: Comparison of Olanzapine and Metoclopramide For Treatment Of bReakThrough Emesis
Acronym: COMFORT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor enrolment
Sponsor: Karin Jordan (Other)
Responsible Party: Sponsor-Investigator, Karin Jordan, MD, Martin-Luther-Universität Halle-Wittenberg
Organization: Martin-Luther-Universität Halle-Wittenberg (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KKSH 079; 2010-018665-30 (EudraCT Number)
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Emesis
Keywords: break-through; emesis; break through emesis after prophylaxis with dexamethasone, 5-HT 3RA and aprepitant
MeSH Terms: conditions — Vomiting | interventions — Olanzapine; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- olanzapine (Experimental)
  Interventions: Drug: olanzapine
- metoclopramide (Active Comparator)
  Interventions: Drug: metoclopramide

INTERVENTIONS:
Drug: olanzapine — 1x10mg per day for three days
  Other Names: Zyprexa
  Arms: olanzapine
Drug: metoclopramide — 3x10mg per day for three days
  Other Names: Paspertin
  Arms: metoclopramide

SUMMARY:
This trial is designed to evaluate olanzapine compared to the metoclopramide in the treatment of break through emesis after prophylaxis with dexamethasone, 5-HT 3 receptor antagonists and aprepitant in patients receiving chemotherapy. Efficacy will be assessed using a modified MASCC questionaire with a visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* break through emesis after prophylaxis with dexamethasone, 5-HT 3 receptor antagonists and aprepitant in patients receiving chemotherapy defined as vomitus or nausea>25mm on VAS
* signed IC

Exclusion Criteria:

* psychiatric disorders
* drug abuse
* pregnancy
* high dose chemotherapy
* treatment with other antiemetic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-07; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate | three days
  no vomitus, no further rescue medication, nausea < 25mm on the visual analog scale (VAS) or reduction on the VAS of >50%

SECONDARY OUTCOMES:
safety | five days
  according to NCI-CTC-AE version4.0
Quality of life | 5 days
  using EORTC-QLQ-C30
change in urinary excretion of 5 hydroxy indole acetic acid | 5 days
  measurement in 24 hours urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Karin Jordan, MD, Principal Investigator — Martin-Luther-University Halle-Wittenberg
Locations (1):
- Martin-Luther-University Halle-Wittenberg, Department for Oncology and Hematology, Ernst-Grube-Strasse 40, Halle, Saxony-Anhalt, Germany